CLINICAL TRIAL: NCT01629667
Title: A Phase 2, Randomized Dose-ranging Study to Evaluate the Efficacy of Tralokinumab in Adults With Idiopathic Pulmonary Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination of the study due to lack of efficacy.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CD-RI-CAT-354-1066
Record Dates: First submitted 2012-06-12; First posted 2012-06-27 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — tralokinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tralokinumab 400 milligram (mg) (Experimental): Participants will receive Tralokinumab 400 mg intravenous (IV) infusion Q4W for 68 Weeks.
  Interventions: Biological: Tralokinumab
- Tralokinumab 800 mg (Experimental): Participants will receive Tralokinumab 800 mg IV infusion Q4W for 68 Weeks.
  Interventions: Biological: Tralokinumab
- Placebo (Placebo Comparator): Participants will receive placebo IV once every 4 Weeks (Q4W) for 68 Weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tralokinumab — Participants will receive Tralokinumab 400 mg IV infusion Q4W for 68 Weeks.
  Arms: Tralokinumab 400 milligram (mg)
Biological: Tralokinumab — Participants will receive Tralokinumab 800 mg IV infusion Q4W for 68 Weeks.
  Arms: Tralokinumab 800 mg
Other: Placebo — Participants will receive placebo IV once every 4 Weeks (Q4W) for 68 Weeks.
  Arms: Placebo

SUMMARY:
To study the safety and effectiveness of multiple-doses of tralokinumab on pulmonary function in adults with mild to moderate idiopathic pulmonary fibrosis (IPF). IPF is a chronic, progressive, irreversible, and usually fatal lung disease of unknown cause.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the effect of multiple doses of tralokinumab on pulmonary function in adults with mild to moderate IPF

ELIGIBILITY:
Key Inclusion Criteria:

* 1) IPF diagnosis for <= 5 years prior to Visit 1 (screening). Confirmation of diagnosis of IPF in accordance is required for subject inclusion 2) Confirmed diagnosis of IPF by clinical characteristics, HRCT and surgical lung biopsy (if required) 3)Mild to moderate IPF to include all of the following at screening:

  1. FVC >= 50% predicted normal
  2. Partial pressure of oxygen in arterial blood (PaO2) of >= 55 mmHg on room air or 50 mmHg at high altitude (> 1500 meters), or oxygen saturation by pulse oximetry (SpO2) of >= 90%on room air at rest
  3. Hemoglobin-corrected diffusion capacity for carbon monoxide (DLCO) >= 30% predicted normal 4) Be able to walk >= 100 meters unassisted

Key Exclusion Criteria:

1. A FEV1/FVC ratio less than 0.70 at the time of screening (postbronchodilator)
2. The extent of emphysema on the HRCT is greater than the extent of fibrosis.
3. Currently listed for lung transplantation
4. Use of the following medications:

   1. Immunosuppressive medications (eg, methotrexate, cyclosporine, azathioprine, intramuscular long-acting depot corticosteroid) within 3 months prior to Visit 1 (screening). Oral prednisone <= 15 mg/day (or equivalent oral corticosteroid) is allowed for chronic use if subject was on a stable dose at least 30 days prior to Visit 1 (screening)
   2. Pirfenidone within 4 weeks prior to Visit 1 (screening)
   3. N-acetylcysteine within 4 weeks prior to Visit 1 (screening)
   4. Live attenuated vaccines within 4 weeks prior to Visit 1 (screening)

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Parker, MD, Study Director — MedImmune LLC
Locations (45):
- United States (21):
  - Research Site, Phoenix, Arizona
  - Research Site, La Jolla, California
  - Research Site, Sacramento, California
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Ann Arbor, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Chesterfield, Missouri
  - Research Site, Summit, New Jersey
  - Research Site, Durham, North Carolina
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, McAllen, Texas
  - Research Site, McKinney, Texas
  - Research Site, Salt Lake City, Utah
- Australia (10):
  - Research Site, Box Hill
  - Research Site, Camperdown
  - Research Site, Concord
  - Research Site, Darlinghurst
  - Research Site, Frankston
  - Research Site, Glen Osmond
  - Research Site, New Lambton
  - Research Site, Parkville
  - Research Site, Prahran
  - Research Site, Woodville South
- Canada (5):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Israel (6):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Rehovot
  - Research Site, Tel Aviv
- Peru (2):
  - Research Site, Lima
  - Research Site, Lima Cercado
- Research Site, Seoul, South Korea

REFERENCES:
- [Derived] Parker JM, Glaspole IN, Lancaster LH, Haddad TJ, She D, Roseti SL, Fiening JP, Grant EP, Kell CM, Flaherty KR. A Phase 2 Randomized Controlled Study of Tralokinumab in Subjects with Idiopathic Pulmonary Fibrosis. Am J Respir Crit Care Med. 2018 Jan 1;197(1):94-103. doi: 10.1164/rccm.201704-0784OC. PMID 28787186

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 409 participants participated in the study. Of which, 176 participants were randomized into the study at 48 sites including 17 sites in the USA, 9 sites in Australia, 7 sites in Peru, 6 sites in Israel, 5 sites in Canada, and 4 sites in South Korea.
Pre-assignment Details: A total of 176 participants were randomized into the study. Three participants who were randomized did not receive treatment; therefore, 173 participants were randomized and treated.
Groups:
- Placebo: Participants received placebo intravenous (IV) once every 4 Weeks (Q4W) for 68 Weeks.
- Tralokinumab 400 Milligram (mg): Participants received Tralokinumab 400 mg IV infusion Q4W for 68 Weeks.
- Tralokinumab 800 mg: Participants received Tralokinumab 800 mg IV infusion Q4W for 68 Weeks.
Period: Overall Study
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Started | 59 | 58 | 59
Randomized and Treated | 57 | 57 | 59
Completed | 12 | 17 | 14
Not Completed | 47 | 41 | 45
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 31 | 20 | 28
Not completed — Death | 1 | 5 | 3
Not completed — Randomized, not treated | 2 | 1 | 0
Not completed — Ongoing AE worsening right heart failure | 0 | 1 | 0
Not completed — Requiring lung transplant | 2 | 1 | 3
Not completed — Early tretmt termntd, cmpltd safety f-up | 9 | 11 | 8
Not completed — Started other medicine | 1 | 0 | 1
Not completed — Site error in safety follow-up | 0 | 0 | 1
Not completed — Enrolled in another clinical study | 0 | 1 | 0
Not completed — Code break | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population is all randomized participants who receive any study investigational product and participants were analysed according to the randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg | Total
Number analyzed (Participants) | 57 | 57 | 59 | 173
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.5 (6.1) | 67.3 (7.7) | 67.9 (6.7) | 67.6 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 13 | 40
  Male | 45 | 42 | 46 | 133

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percent-predicted Forced Vital Capacity (FVC) at Week 52
Description: Forced vital capacity (FVC) is a standard pulmonary function test used to monitor disease progression in IPF. FVC was the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in litres. Predicted forced vital capacity is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FVC = (observed value)/(predicted value) * 100%.
Time Frame: Baseline and Week 52
Population: The intent-to-treat (ITT) population included all randomized participants who received any study investigational product and participants were analysed according to the randomization. Here, "n" is number of participants analysed at given time point.
Measure: Mean (Standard Deviation); unit: Percentage of predicted FVC
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Percentage of predicted FVC
  Baseline (n=57,57,59) | 70.30 (12.04) | 68.54 (14.26) | 70.60 (13.37)
  Change at Week 52 (n=36,32,35) | -4.08 (6.85) | -6.10 (6.98) | -6.07 (5.14)
Statistical Analysis 1: Comparison: Placebo vs Tralokinumab 400 Milligram (mg); Test type: Superiority or Other; p = 0.140, ANCOVA; Least square mean difference = -1.77, 95% CI 2-sided [-4.13 to 0.59]
Statistical Analysis 2: Comparison: Placebo vs Tralokinumab 800 mg; Test type: Superiority or Other; p = 0.234, ANCOVA; Least square mean difference = -1.41, 95% CI 2-sided [-3.73 to 0.91]

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: Any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening situation (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received Tralokinumab. Treatment-emergent were events between administration of investigational product and Week 88 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the start of study treatment through Week 88
Population: The safety population included all participants who received any study investigational product and participants were analysed according to the treatment they actually received.
Measure: Number; unit: Participant
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Participant
  TEAE | 53 | 50 | 57
  TESAE | 13 | 16 | 17

3. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as Treatment-emergent Adverse Events
Description: An abnormal laboratory finding which required an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation were reported as an adverse event. Treatment-emergent were events between administration of investigational product and Week 88 that were absent before treatment or that worsened relative to pre-treatment state. Laboratory evaluations (haematology, serum chemistry and urinalysis) of blood and urine samples were performed.
Time Frame: From the start of study treatment through Week 88
Population: as for outcome 2
Measure: Number; unit: Participant
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Participant
  Anaemia | 1 | 0 | 1
  Haemoglobin decreased | 0 | 1 | 0
  Hypovolaemia | 1 | 0 | 0
  ALT increased | 0 | 0 | 1
  AST increased | 0 | 0 | 1
  Blood glucose increased | 0 | 0 | 1
  Diabetes mellitus | 2 | 0 | 0
  Diabetes mellitus inadequate control | 0 | 1 | 0
  Type 2 diabetes mellitus | 0 | 0 | 1
  Gout | 0 | 1 | 1
  Hepatic steatosis | 0 | 0 | 1
  Liver function test abnormal | 0 | 0 | 1
  GGT increased | 0 | 0 | 1
  Hyperlipidaemia | 0 | 0 | 1
  Hyperglycaemia | 1 | 0 | 0
  Hypokalaemia | 1 | 0 | 0
  Hypertriglyceridaemia | 1 | 0 | 0
  Hyponatraemia | 1 | 0 | 0
  Hypophosphataemia | 0 | 0 | 1
  Iron deficiency | 1 | 0 | 0
  Vitamin D deficiency | 0 | 1 | 0
  Vitamin D decreased | 0 | 0 | 1

4. Secondary Outcome: Number of Participants With Vital Signs and Physical Findings Abnormalities Reported as Treatment-emergent Adverse Events
Description: Vital signs parameters included heart rate, blood pressure, temperature, weight, pulse oximetry and respiratory rate. Treatment-emergent were events between administration of investigational product and Week 88 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: From the start of study treatment through Week 88
Population: as for outcome 2
Measure: Number; unit: Participant
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Participant
  Hypertension | 2 | 1 | 2
  Pulmonary hypertension | 2 | 1 | 2
  Pyrexia | 1 | 1 | 2
  Hypotension | 1 | 1 | 1
  Blood pressure increased | 0 | 0 | 2
  Atrial fibrillation | 0 | 0 | 2
  Atrial flutter | 1 | 0 | 1
  Arrhythmia | 0 | 0 | 1
  Bradycardia | 1 | 0 | 0
  Heart rate increased | 0 | 0 | 1
  Palpitations | 0 | 0 | 1
  Sinus tachycardia | 1 | 0 | 0
  Supraventricular tachycardia | 1 | 0 | 0
  Tachyarrhythmia | 0 | 0 | 1
  Weight decreased | 4 | 5 | 3

5. Secondary Outcome: Number of Participants With Electrocardiogram Abnormalities Reported as Treatment-emergent Adverse Events
Description: AEs observed in participants with clinically significant ECG abnormalities were assessed. Tricuspid valve incompetence was the only abnormality reported as TEAE. ECG parameters included heart rate, PR, QRS, QT, and QTc intervals. Treatment-emergent were events between administration of investigational product and Week 88 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: From the start of study treatment through Week 88
Population: as for outcome 2
Measure: Number; unit: Participant
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Participant | 1 | 0 | 1

6. Secondary Outcome: Percentage of Participants With Disease Progression
Description: Progression-free Survival (PFS) was used to evaluate disease progression and the percentage of participants with disease progression. A participant was classified as having disease progression if at least one of the following criteria were met:• Adjudicated respiratory-related mortality. •Adjudicated hospitalization due to IPF exacerbation. •Confirmed decline in percent-predicted FVC of greater than or equal to (>=) 10%. •Confirmed decline in 6 minute walk test (6MWT) >= 50 meters.
Time Frame: Week 52 and 72
Population: The intent-to-treat (ITT) population included all randomized participants who received any study investigational product and participants were analysed according to the randomization.
Measure: Number; unit: Percentage of Participant
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Percentage of Participant
  At Week 52 | 35.1 | 35.1 | 28.8
  At Week 72 | 42.1 | 42.1 | 44.1

7. Secondary Outcome: Change From Baseline in Haemoglobin (Hb) Corrected Percent-predicted Diffusion Capacity for Carbon Monoxide (DLco) Through Week 72
Description: The single breath technique was used to determine the DLco. The test was performed by qualified pulmonary function technicians with experience performing this study. Acceptable test criteria included:• An inspiratory volume of more than 85% of vital capacity. • A stable breath hold of 10 seconds (+/- 2 seconds) with no leaks, Valsalva or Mueller maneuvers. • Expiration in less than 4 seconds with appropriate clearance of dead space. The average of the two best acceptable maneuvers was used. There must be a minimum of 4 minutes between the performances of each test.
Time Frame: Baseline, Week 52 and 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent predicted DLco
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Percent predicted DLco
  Baseline (n=57,57,59) | 46.962 (13.796) | 49.389 (16.029) | 47.509 (12.524)
  Change at Week 52 (n=34,30,32) | -3.963 (8.777) | -5.233 (9.597) | -6.356 (8.588)
  Change at Week 72 (n=23,21,22) | -8.322 (9.538) | -9.962 (10.362) | -10.382 (12.372)

8. Secondary Outcome: Change From Baseline in 6 Minute Walk Test (6MWT) Distance Through Week 72
Description: The 6MWT measures the distance that a participant can walk on a measured, flat hard surface in a period of 6 minutes. The 6MWT evaluates the global and integrated responses of all body systems involved during walking.
Time Frame: Baseline, Week 52 and 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Meter
  Baseline (n=55,57,56) | 391.07 (112.06) | 391.69 (102.46) | 383.22 (93.99)
  Change at Week 52 (n=31,31,29) | 19.49 (71.36) | 22.96 (52.38) | -12.40 (55.81)
  Change at Week 72 (n=21,24,19) | 18.76 (54.83) | 7.85 (78.12) | -30.25 (78.07)

9. Secondary Outcome: Change From Baseline in Oxygen Saturation by Pulse Oximetry at Week 68
Description: Participants transcutaneous oxygen saturation were observed by pulse oximetry.
Time Frame: Baseline and Week 68
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of oxygen saturation
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Percent of oxygen saturation
  Baseline (n=57,57,59) | 96.2 (1.9) | 95.6 (2.0) | 95.4 (2.9)
  Change at Week 52 (n=30,28,29) | -0.6 (2.3) | 0.4 (1.7) | -0.7 (2.7)
  Change at Week 68 (n=23,25,22) | -0.6 (1.8) | 0.1 (2.4) | -1.0 (2.8)

10. Secondary Outcome: Change From Baseline in Lung Volumes Through Week 72
Description: Lung volumes were evaluated by total lung capacity (TLC), residual volume (RV), and vital capacity (VC). Lung volumes were determined by body plethysmography.
Time Frame: Baseline, Week 52 and 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Liter
  Baseline (n=53,50,53) | 4.105 (0.905) | 3.870 (0.905) | 4.060 (1.192)
  Change at Week 52 (n=32,29,28) | 0.891 (5.150) | -0.212 (0.645) | -0.264 (0.442)
  Change at Week 72 (n=24,22,19) | -0.139 (0.635) | -0.274 (0.705) | -0.417 (0.468)

11. Secondary Outcome: Percentage of Participants With Idiopathic Pulmonary Fibrosis (IPF) Exacerbations
Description: The IPF exacerbations is defined as an acute, clinically significant, deterioration of unidentifiable cause in a participant with underlying IPF. Exacerbations of IPF were adjudicated according to the protocol definition by an independent committee as follows:
  1. Confirmed acute IPF exacerbation, 2. Suspected acute IPF exacerbation, 3. Not an IPF exacerbation with an alternative diagnosis provided if possible, and 4. Undetermined due to insufficient information.
Time Frame: Week 52 and 72
Population: as for outcome 6
Measure: Number; unit: Percentage of participant
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Percentage of participant
  At Week 52 | 12.3 | 12.3 | 8.5
  At Week 72 | 12.3 | 17.5 | 11.9

12. Secondary Outcome: Percentage of Participants With Adjudicated Mortality
Description: Participants all cause mortality were observed. Events that resulted in participant death were adjudicated into respiratory-related mortality or all other cause mortality by an independent committee.
Time Frame: Week 52 and 72
Population: as for outcome 6
Measure: Number; unit: Percentage of participant
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Percentage of participant
  At Week 52 | 3.5 | 7.0 | 5.1
  At Week 72 | 3.5 | 8.8 | 5.1

13. Secondary Outcome: Percentage of Participants With Adjudicated Hospitalization
Description: Participants who were hospitalized due to IPF exacerbation were observed. All events that resulted in the hospitalization of participants were adjudicated by an independent committee to determine if the event was due to an IPF exacerbation as follows: 1. Exacerbation or progression of IPF, 2. Result of a complication of IPF, 3. Not related to IPF (alternative diagnosis provided), and 4. Undetermined due to insufficient information.
Time Frame: Week 52 and 72
Population: as for outcome 6
Measure: Number; unit: Percentage of participant
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Percentage of participant
  At Week 52 | 21.1 | 24.6 | 16.9
  At Week 72 | 21.1 | 24.6 | 23.7

14. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Through Week 72
Description: FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration.
Time Frame: Baseline, Week 52 and 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Liter
  Baseline (n=57,57,59) | 2.199 (0.500) | 2.025 (0.495) | 2.144 (0.564)
  Change at Week 52 (n=36,32,35) | -0.120 (0.259) | -0.148 (0.200) | -0.179 (0.134)
  Change at Week 72 (n=26,26,23) | -0.260 (0.261) | -0.152 (0.317) | -0.222 (0.166)

15. Secondary Outcome: Change From Baseline in Percent-predicted FEV1 Through Week 72
Description: FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Predicted FEV1 is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FEV1 = (observed value)/(predicted value) * 100%.
Time Frame: Baseline, Week 52 and 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of predicted FEV1
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Percent of predicted FEV1
  Baseline (n=57,57,59) | 78.56 (13.05) | 77.88 (14.88) | 78.94 (14.58)
  Change at Week 52 (n=36,32,35) | -4.16 (8.50) | -5.78 (8.11) | -7.01 (5.33)
  Change at Week 72 (n=26,26,23) | -8.77 (8.99) | -6.42 (11.13) | -8.61 (6.61)

16. Secondary Outcome: Change From Baseline in Absolute Forced Vital Capacity (FVC) Through Week 72
Description: Forced vital capacity (FVC) is a standard pulmonary function test used to monitor disease progression in IPF. FVC was the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in litres.
Time Frame: Baseline, Week 52 and 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Liter
  Baseline (n=57,57,59) | 2.662 (0.649) | 2.406 (0.664) | 2.593 (0.711)
  Change at Week 52 (n=36,32,35) | -0.162 (0.278) | -0.205 (0.224) | -0.209 (0.168)
  Change at Week 72 (n=26,26,23) | -0.322 (0.297) | -0.186 (0.325) | -0.282 (0.242)

17. Secondary Outcome: Number of Participants With Clinical Global Impression of Severity Scores
Description: The CGI-S is a single, clinician completed, item designed to capture the clinician's impression of the participants IPF severity. Clinicians were asked to consider their experience in this participant population and rate the overall IPF severity of the participant using a 5-point scale (1 = very mild, 5 = very severe).
Time Frame: Week 72
Population: The intent-to-treat (ITT) population included all randomized participants who received any study investigational product and participants were analysed according to the randomization. Here, "N" is number of participants analysed for this outcome measure.
Measure: Number; unit: Participant
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 25 | 24 | 24
Participant
  Very mild | 1 | 0 | 1
  Mild | 6 | 10 | 6
  Moderate | 16 | 10 | 11
  Severe | 0 | 3 | 5
  Very severe | 2 | 1 | 1

18. Secondary Outcome: Number of Participants With Clinical Global Impression of Change Scores
Description: The CGI-C is a single, clinician completed, item designed to capture the clinicians overall impression of change in IPF severity from the baseline state at Screening. Clinicians were asked to rate the participants IPF severity relative to their state at baseline using a 7-point scale (-3 = very much worse, 0 = no change, about the same, 3 = very much improved).
Time Frame: Week 72
Population: as for outcome 17
Measure: Number; unit: Participant
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 25 | 24 | 23
Participant
  Very much improved | 0 | 0 | 0
  Much improved | 1 | 0 | 3
  Slightly improved | 2 | 1 | 1
  No change | 12 | 13 | 8
  Slightly worse | 8 | 8 | 6
  Much worse | 1 | 2 | 4
  Very much worse | 1 | 0 | 1

19. Secondary Outcome: Change From Baseline in University of California San Diego Shortness of Breath Questionnaire (UCSD SOBQ) Total Score at Week 72
Description: The UCSD SOBQ is a 24-item questionnaire designed to capture patient-reported shortness of breath. Respondents were asked to rate their breathlessness during 21 activities of daily living using a 6-point scale (0 = not at all breathless, 5 = maximally breathless or too breathless to do this activity). In addition to the 21 activity items, the UCSD SOBQ includes 3 additional questions about limitations due to shortness of breath, fear of harm from overexertion, and fear of shortness of breath. The UCSD SOBQ was scored by summing responses across all 24 items to form a total score. Scores range from 0-120 with higher scores indicative of greater shortness of breath.
Time Frame: Baseline and Week 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Units on a scale
  Baseline (n=56,55,58) | 40.9 (22.8) | 36.5 (21.0) | 45.9 (20.4)
  Change at Week 72 (n=24,21,21) | 12.9 (14.7) | -0.4 (18.0) | 10.9 (23.3)

20. Secondary Outcome: Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score at Week 72
Description: The SGRQ is a 50-item Patient-reported outcome (PRO) instrument developed to measure respiratory-related health status via 76 weighted responses. The SGRQ is divided into two parts. Part 1 asks respondents to consider the last 3 months and report on their respiratory symptoms using 5-point Likert scales. Part 2 asks respondents to consider their current state and respond to a series of dichotomous yes/no items related to their activities (activities that cause or were limited by breathlessness) and impacts (social functioning, psychological disturbances resulting from airways disease). Total scores and domain scores (symptoms, activities, and impact on daily life) were scored from 0-100, where lower scores indicate better health status.
Time Frame: Baseline and Week 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Units on a scale
  Baseline (n=57,57,59) | 47.24 (18.86) | 44.80 (18.91) | 51.39 (15.64)
  Change at Week 72 (n=24,24,23) | 2.91 (14.92) | 3.16 (15.11) | 3.38 (14.88)

21. Secondary Outcome: Change From Baseline in Exacerbations of Chronic Pulmonary Disease (EXACT IPF) Total Score Through Week 72
Description: The EXACT-IPF is a 14-item daily dairy used to capture the IPF related symptoms completed by the participants using an eDiary. The EXACT-IPF total score is the sum of all items ranged from 1 to 14. EXACT-IPF is an interval-level scale ranging from 0 to 100, where the higher scores indicate more severe condition. The EXACT-IPF used Likert scales (with 3 to 6 response options each) to capture participant reported IPF-related symptoms. The scores are the simple sum of item responses for each domain or single item.
Time Frame: Baseline, Week 52 and 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Units on a scale
  Baseline (n=55,51,56) | 16.24 (9.44) | 15.87 (8.38) | 17.89 (9.72)
  Change at Week 52 (n=31,27,30) | 1.47 (5.75) | 1.61 (7.21) | 1.40 (10.18)
  Change at Week 72 (n=23,23,20) | 1.95 (7.46) | 0.63 (7.50) | 1.81 (10.00)

22. Secondary Outcome: Change From Baseline in European Quality of Life-5-Dimension 3 Level Version (EQ-5D-3L) (Including Visual Analog Scale [VAS]) at Week 72
Description: The EQ-5D-3L is a standardized PRO used to capture respondent's general health status. The questionnaire assesses 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 response options (no problem, some or moderate problems, and unable or extreme problems) that reflect increasing levels of difficulty. The questionnaire also includes a visual analog scale, where the participants were asked to rate their current health on a scale of 0-100, with 0 being the worst imaginable health state.
Time Frame: Baseline and Week 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Units on a scale
  Baseline (n=57,57,59) | 70.5 (19.1) | 70.5 (18.1) | 66.6 (14.9)
  Change at Week 72 (n=24,24,23) | -3.0 (17.9) | 2.5 (20.9) | 0.6 (14.3)

23. Secondary Outcome: Number of Participants With Patient Global Impression of Severity (PGI-S) for Idiopathic Pulmonary Fibrosis (IPF)
Description: The PGI-S is a single-item, global assessment of participant-perceived IPF severity. The assessment was designed to capture participant perceived IPF-related health status. Participants rate their IPF severity using a 5-point scale (1 = very mild, 5 = very severe).
Time Frame: Week 72
Population: as for outcome 17
Measure: Number; unit: Participant
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 23 | 21 | 15
Participant
  Very mild | 2 | 2 | 1
  Mild | 8 | 5 | 6
  Moderate | 11 | 13 | 8
  Severe | 1 | 1 | 0
  Very severe | 1 | 0 | 0

24. Secondary Outcome: Number of Participants With Patient Global Impression of Change (PGI-C) for Idiopathic Pulmonary Fibrosis (IPF)
Description: The PGI-C is a single-item, global assessment designed to capture participant-perceived change in their IPF health condition using a 7-point scale (-3 = very much improved, 0 = no change, about the same, 3 = very much worse).
Time Frame: Week 72
Population: as for outcome 17
Measure: Number; unit: Participant
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 7 | 11 | 14
Participant
  Very much improved | 0 | 0 | 0
  Much improved | 1 | 1 | 0
  Slightly improved | 1 | 4 | 4
  No change | 1 | 3 | 5
  Slightly worse | 3 | 2 | 3
  Much worse | 1 | 1 | 2
  Very much worse | 0 | 0 | 0

25. Secondary Outcome: Mean Serum Concentration of Tralokinumab
Description: The mean serum concentration of Tralokinumab were observed.
Time Frame: Predose, 0 hour, and 2 hour postdose on Week 0; predose on Week 4, 48, 72, 82 and 88
Population: The Pharmacokinetic population included all participants who received at least one dose of tralokinumab and had at least one detectable trough (Weeks 4, 48 or 72 only) serum concentration measurement. Here, "n" is number of participants analysed at given time point.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/ml)
Arm/Group | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 59
microgram per milliliter (mcg/ml)
  Week 0: predose (n=50,56) | 3.520 (23.885) | 6.151 (45.560)
  Week 0: 0 hour postdose (n=53,57) | 176.047 (125.991) | 311.105 (88.229)
  Week 0: 2 hour postdose (n=53,56) | 172.108 (46.423) | 301.321 (60.520)
  Week 4 (n=57,57) | 30.155 (20.164) | 57.914 (45.326)
  Week 48 (n=33,39) | 44.653 (40.584) | 80.553 (67.187)
  Week 72 (n=24,21) | 41.583 (24.723) | 76.224 (54.045)
  Week 82 (n=15,12) | 3.651 (3.547) | 11.442 (13.846)
  Week 88 (n=12,10) | 0.493 (0.490) | 10.585 (19.084)

26. Secondary Outcome: Percentage of Participants Positive for Anti-Drug Antibodies to Tralokinumab
Description: A participant was considered ADA-positive across the study if they had a positive reading at any time point during the study.
Time Frame: From the start of study treatment through Week 88
Population: The safety population included all participants who received any study investigational product and participants were analysed according to the treatment they actually received. Here, "n" is number of participants analysed at given time point.
Measure: Number; unit: Percentage of participant
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Number analyzed (Participants) | 57 | 57 | 59
Percentage of participant
  Baseline (n=54,54,58) | 1.9 | 1.9 | 0
  Week 0, Day 1 (n=1,3,1) | 0 | 0 | 0
  Week 48 (n=35,32,36) | 2.9 | 0 | 0
  Week 72 (n=2,1,1) | 0 | 0 | 0
  Week 82 (n=13,15,12) | 7.7 | 0 | 0
  Week 88 (n=10,13,11) | 20 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of study treatment through Week 88 or at the time of early termination from the study
Arm/Group | Placebo | Tralokinumab 400 Milligram (mg) | Tralokinumab 800 mg
Serious Adverse Events (participants affected / at risk) | 13/57 | 16/57 | 17/59
Other Adverse Events (participants affected / at risk) | 51/57 | 45/57 | 50/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=57) | Tralokinumab 400 Milligram (mg) (N=57) | Tralokinumab 800 mg (N=59)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Appendiceal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 6 (7) | 2 (2)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (4) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 7 (7) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=57) | Tralokinumab 400 Milligram (mg) (N=57) | Tralokinumab 800 mg (N=59)
Constipation (Gastrointestinal disorders) | 4 (6) | 3 (6) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 6 (10) | 4 (5) | 9 (20)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (19) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (7) | 6 (9)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (1) | 3 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 4 (4)
Fatigue (General disorders) | 4 (4) | 5 (22) | 11 (11)
Oedema peripheral (General disorders) | 4 (5) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 1 (2) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 5 (7) | 7 (9) | 5 (8)
Herpes zoster (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 4 (5) | 3 (3) | 5 (8)
Nasopharyngitis (Infections and infestations) | 6 (6) | 6 (9) | 5 (8)
Pharyngitis (Infections and infestations) | 2 (2) | 6 (7) | 3 (3)
Respiratory tract infection (Infections and infestations) | 4 (5) | 1 (1) | 3 (7)
Sinusitis (Infections and infestations) | 6 (7) | 1 (6) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 7 (16) | 10 (20) | 11 (14)
Urinary tract infection (Infections and infestations) | 3 (5) | 3 (3) | 4 (5)
Viral upper respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 4 (7)
Laceration (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 4 (4) | 5 (6) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (9) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (6) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3) | 6 (6)
Headache (Nervous system disorders) | 8 (12) | 6 (12) | 5 (9)
Lethargy (Nervous system disorders) | 2 (2) | 2 (3) | 1 (1)
Syncope (Nervous system disorders) | 2 (3) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (4) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 8 (9) | 2 (2) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 10 (12) | 17 (28)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (12) | 10 (14)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (2)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 8 (8) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 5 (9)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (3) | 5 (5)
Haematoma (Vascular disorders) | 0 (0) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Study was early terminated due to lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.